CLINICAL TRIAL: NCT00205205
Title: Peer Mentoring for Persons With Spinal Cord Injury: Program Satisfaction and Outcome for Mentor/Mentee
Brief Title: Peer Mentoring for Persons With Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2003-0505
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-06

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Behavioral: peer mentoring

SUMMARY:
A peer mentoring program for persons with SCI was developed. Individuals who experienced SCI in the past and have adapted well functionally were asked to serve as mentors for individuals with newly-acquired SCI. These individuals undergo volunteer and peer mentoring training prior to mentoring activities. They are a subset of the study participants. We are tracking their satisfaction with life, positive and negative affect, life adjustment, depression, and social support over time. We hypothesize that measures of adjustment will become more positive as involvement as a mentor increases. The second subset of study participants are the individuals with newly-acquired SCI. They complete a baseline assessment of the measures listed above and then at 6 months, one year, and two years after match with a mentor. We also collect information about the quantity and quality of the mentoring sessions from both the mentor and mentee. We hypothesize that the mentee's adjustment will be positively influenced by the number and quality of the mentoring sessions. Due to the relatively small number of SCI per year in our program, we opted to offer the mentoring program to all individuals with newly acquired SCI, thus there is no control group.

ELIGIBILITY:
Inclusion Criteria:

* experienced a SCI

Exclusion Criteria:

* no severe traumatic brain injury
* no severe psychiatric disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
satisfaction with life, positive and negative affect, life adjustment, depression, and social support

SECONDARY OUTCOMES:
is the mentee's adjustment positively influenced by the number and quality of the mentoring sessions

CONTACTS AND LOCATIONS:
Overall Officials: Jack Sherman, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Veith, E.M., Sherman, J.E., Pellino, T.A. Yasui, T.Y. (2006). Qualitative analysis of the peer-mentoring relationship among individuals with spinal cord injury, Rehabilitation Psychology, 51, 289-298.